CLINICAL TRIAL: NCT01236495
Title: Comparison for Pethidine Requirement in Patients Received Spinal Morphine 0.2 and 0.3 Milligram for Post Lobectomy (Lung) Analgesia
Brief Title: Comparison for Pethidine Requirement in Patients Received Spinal Morphine 0.2 and 0.3 mg for Post Lobectomy Analgesia
Acronym: pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: si578/2010
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Solitary Mass; Lung Diseases
Keywords: thoracotomy; postoperative pain; spinal morphine
MeSH Terms: conditions — Lung Diseases; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal morphine 0.2 mg (Experimental): spinal morphine 0.2 mg
  Interventions: Drug: spinal morphine 0.2 mg
- spinal morphine 0.3 mg (Active Comparator): spinal morphine 0.3 mg
  Interventions: Drug: spinal morphine 0.3 mg

INTERVENTIONS:
Drug: spinal morphine 0.3 mg — spinal morphine 0.3 mg
  Other Names: morphine
  Arms: spinal morphine 0.3 mg
Drug: spinal morphine 0.2 mg — spinal morphine 0.2 mg
  Other Names: morphine
  Arms: spinal morphine 0.2 mg

SUMMARY:
The purpose of the study is to evaluate the amount of total pethidine requirement during the 48 hour postoperative period after receiving spinal morphine 0.2 and 0.3 mg.

DETAILED DESCRIPTION:
Thoracotomy causes severe pain to the patients. Continuous thoracic epidural is a gold standard for postoperative pain. However, it needs skill. There are many alternatives such as spinal morphine, intercostal nerve block, cryoalangesia or interpleural block.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year and < 70 year
* Patient ASA physical status I-III.
* Scheduled for thoracotomy with lobectomy.
* Can operate a patient-controlled analgesia (PCA) device.

Exclusion Criteria:

* Known hypersensitivity to morphine or pethidine
* History of bleeding tendency.
* Known case of infection at the back
* Patient refuse for spinal anesthesia
* History of cerebrovascular disease.
* Scheduled for video-assisted thoracoscopic lobectomy.
* Need mechanical ventilatory support during postoperative period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
pethidine requirement | 48 hours
  Total pethidine requirement during 48 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, M.D., Principal Investigator — Deaprt ment of Anesthesiology ,Faculty of Medicine, Siriraj Hospital
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand